CLINICAL TRIAL: NCT03087851
Title: Treatment With Zoledronic Acid Subsequent to Denosumab in Osteoporosis
Acronym: ZOLARMAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Anne Sophie Sølling, MD, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-005529-37
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Osteoporosis
Keywords: Denosumab; Bone turnover markers; Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 6-month group (Active Comparator): Zoledronic acid will be administered at study day 0. If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site a second infusion of zoledronic acid will be administered.
  Interventions: Drug: Zoledronic Acid
- 9-months group (Active Comparator): Zoledronic acid will be administered depending on increase in s-CTX (above 1.26 ug/l) or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 3.
  If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site a second infusion of zoledronic acid will be administered.
  Interventions: Drug: Zoledronic Acid
- Observation group (Active Comparator): Zoledronic acid will be administered depending on increase in s-CTX (above 1.26 ug/l), decrease in BMD (more than 5% at any site), or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 6.
  If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site a second infusion of zoledronic acid will be administered.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Intravenous infusion of 5 mg zoledronic acid
  Other Names: Zoledronate

SUMMARY:
Denosumab is an antibody against receptor-activator of nuclear factor kappa-B ligand that prevents recruitment and differentiation of mature osteoclasts. Treatment markedly decrease bone resorption and fracture risk, and many patients will reach osteopenic bone mineral density (BMD) levels on treatment with denosumab. The treatment effect on bone turnover and BMD has, however, been demonstrated to be reversible. This study will show if the bone mass can be maintained by administrating zoledronic acid and if timing of the first dose of zoledronic acid after last dose of denosumab matters.

DETAILED DESCRIPTION:
Background: Denosumab is an antibody against receptor-activator of nuclear factor kappa-B ligand that prevents recruitment and differentiation of osteoclasts. Treatment decreases bone resorption and fracture risk. After discontinuation, however, bone resorption increases and the bone mass gained during 2 years of therapy is lost within 1 year. At present denosumab treatment is considered to be life-long.

Aim: To investigate if infusion of zoledronic acid can prevent increases in bone turnover and bone loss in patients previously treated with denosumab and if there is difference between infusing zoledronic acid at six or nine months after the last injection of denosumab or when bone turnover is increased.

Methods: A randomized open label, interventional study in 60 patients investigating if treatment with zoledronic acid prevents bone loss after denosumab treatment when administrated six or nine months after last injection of deno-sumab or when bone turnover is increased. Forty patients will be allocated to the two intervention groups and 20 patients will be followed without treatment for up to 12 months after the last denosumab treatment. The patients in the observation group and the nine months group will be monitored monthly and if s-carboxy-terminal collagen cross-links (s-CTX) increases above 1.26ug/l (50% above the normal range for postmenopausal women and elderly men) infusion of zoledronic acid will be administered. Furthermore, a DXA scan (lumbar spine and hip sites) will be performed after three months in the observation group. If BMD has decreased more than 5% at any site, infusion of zoledronic acid will be administered. Finally, if a patient in the 9 months group or the in the observation group suffers an osteoporotic clinical vertebral or hip fracture, infusion of zoledronic acid will be administered.

The patients will be monitored with DXA 6, 12 and 24 months after the infusion of zoledronic acid. Zoledronic acid will be re-administered if BMD has decreased more than 5% at the lumbar spine, total hip or femoral neck. If s-CTX in-creases above 1.26 ug/l during the 2nd year a second infusion of zoledronic acid will be administered.

Perspectives: Many patients will reach osteopenic BMD levels on treatment with denosumab, however the treatment effect on bone turnover and BMD has been demonstrated to be reversible and it is therefore important to find out if denosumab treatment can be discontinued and bone mass maintained by other measures. This study will show if the bone mass can be maintained by administrating zoledronic acid and if timing of the first dose of zoledronic acid after last dose of denosumab matters. If bone loss can be prevented by zoledronic acid expenses on otherwise life-long denosumab treatment can be saved and long-term side effects of denosumab (atypical femur fractures and osteone-crosis of the jaw) can be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal for at least two years)
* Men above 50 years
* Treatment for at least two years with denosumab
* Last denosumab injection less than five months ago

Exclusion Criteria:

* Low-energy vertebral fracture at any time
* Low-energy hip fracture within the last 12 months
* BMD T-score < -2,5 (lumbar spine, total hip or femoral neck)
* Alendronate treatment for more than three years prior to denosumab treatment
* Ongoing treatment with glucocorticoids
* Metabolic bone disease
* Hormone replacement therapy
* Cancer
* Estimated glomerular filtration rate (eGFR) < 35 mL/min
* Allergy to zoledronic acid
* Hypocalcaemia
* Contraindications for zoledronic acid according to the SPC

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bente L Langdahl, MD PhD DMSc, Study Director — Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacey DL, Boyle WJ, Simonet WS, Kostenuik PJ, Dougall WC, Sullivan JK, San Martin J, Dansey R. Bench to bedside: elucidation of the OPG-RANK-RANKL pathway and the development of denosumab. Nat Rev Drug Discov. 2012 May;11(5):401-19. doi: 10.1038/nrd3705. PMID 22543469
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Koldkjaer Solling AS, Harslof T, Kaal A, Rejnmark L, Langdahl B. Hypercalcemia after discontinuation of long-term denosumab treatment. Osteoporos Int. 2016 Jul;27(7):2383-2386. doi: 10.1007/s00198-016-3535-5. Epub 2016 Apr 20. PMID 27098536
- [Background] Aubry-Rozier B, Gonzalez-Rodriguez E, Stoll D, Lamy O. Severe spontaneous vertebral fractures after denosumab discontinuation: three case reports. Osteoporos Int. 2016 May;27(5):1923-5. doi: 10.1007/s00198-015-3380-y. Epub 2015 Oct 28. PMID 26510845
- [Background] Anastasilakis AD, Makras P. Multiple clinical vertebral fractures following denosumab discontinuation. Osteoporos Int. 2016 May;27(5):1929-30. doi: 10.1007/s00198-015-3459-5. Epub 2015 Dec 22. No abstract available. PMID 26694593
- [Background] Shane E, Burr D, Ebeling PR, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster D, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Koval K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Sen HT, van der Meulen MC, Weinstein RS, Whyte M; American Society for Bone and Mineral Research. Atypical subtrochanteric and diaphyseal femoral fractures: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2010 Nov;25(11):2267-94. doi: 10.1002/jbmr.253. PMID 20842676
- [Derived] Solling AS, Harslof T, Langdahl B. Treatment With Zoledronate Subsequent to Denosumab in Osteoporosis: A 2-Year Randomized Study. J Bone Miner Res. 2021 Jul;36(7):1245-1254. doi: 10.1002/jbmr.4305. Epub 2021 Apr 20. PMID 33813753
- [Derived] Solling AS, Harslof T, Langdahl B. Treatment with Zoledronate Subsequent to Denosumab in Osteoporosis: a Randomized Trial. J Bone Miner Res. 2020 Oct;35(10):1858-1870. doi: 10.1002/jbmr.4098. Epub 2020 Jul 12. PMID 32459005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants from the Department of Endocrinology, Aarhus University Hospital, Denmark and via advertisements in newspapers and online. The Danish Health Data Authority provided two data extractions, with information on patients living in the Central Region of Denmark, who had redeemed a minimum of 5 prescriptions for denosumab (DMAB) within the last 3 years.
Groups:
- 6-month Group: Zoledronate: administrated at baseline.
  Zoledronate re-adminisrated:
  If p-C-terminal telopeptide of type 1 collagen (p-CTX) increases above 1.26 ug/l or bone mineral density (BMD) decreases more than 5% at any site.
- 9-months Group: Zoledronate: administrated depending on increase in p-CTX (above 1.26 ug/l) or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 3.
  Zoledronate re-administrated:
  If p-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site.
- Observation Group: Zoledronate: administrated depending on increase in p-CTX (above 1.26 ug/l), decrease in BMD (more than 5%), or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 6.
  Zoledronate re-administrated:
  If p-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site.
Period: Overall Study
Arm/Group | 6-month Group | 9-months Group | Observation Group
Started | 20 | 20 | 21
Completed | 20 | 19 | 19
Not Completed | 0 | 1 | 2
Not completed — Withdraw on medical grounds | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- 6-month Group; 9-months Group; Observation Group: Treated with zoledronate 5 mg
- Total: Total of all reporting groups
Arm/Group | 6-month Group | 9-months Group | Observation Group | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 7 | 27
  >=65 years | 12 | 8 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8) | 65 (7) | 69 (9) | 68 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 19 | 54
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 21 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Lumbar spine BMD [Mean (Standard Deviation); unit: g/cm^2] | 0,880 (0.055) | 0,878 (0,063) | 0,871 (0,089) | 0,876 (0,069)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine BMD From Baseline to 6 Months After the Zoledronic Acid Infusion.
Description: Change in lumbar spine BMD from baseline to 6 months after the zoledronic acid infusion.
Time Frame: baseline to 6 months after the zoledronic acid infusion
Population: Change in lumbar spine BMD from baseline to 6 months after the zoledronic acid infusion.
Measure: Mean (Standard Error); unit: percentage change
Groups:
- 6-month Group; 9-months Group: n=20
- Observation Group: n=21
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
percentage change | -2.1 (0.9) | -4.3 (1.1) | -3.0 (1.1)

2. Primary Outcome: Number of Participants Who Fail to Maintain BMD
Description: Failure is defined as ≥ 3 % BMD loss at the lumbar spine
Time Frame: 2 years after the first ZOL treatment
Population: Number of Participants Who Fail to Maintain lumbar spine BMD from baseline to 24 months after the first ZOL
Measure: Number; unit: participants
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
participants | 10 | 5 | 6

3. Secondary Outcome: Changes in BMD From Baseline to One Year After the Zoledronic Acid Infusion.
Description: Changes in lumbar spine BMD from baseline to one year after the zoledronic acid infusion.
Time Frame: from baseline to one year after the zoledronic acid infusion
Population: Changes in lumbar spine BMD from baseline to one year after the zoledronic acid infusion.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
percentage change | -4.8 (0.7) | -4.1 (1.1) | -4.7 (1.2)

4. Secondary Outcome: Changes in BMD From Baseline to Two Years After the Zoledronic Acid Infusion.
Description: Changes in lumbar spine BMD from baseline to two years after the zoledronic acid infusion.
Time Frame: from baseline to two years after the zoledronic acid infusion.
Population: Changes in lumbar spine BMD from baseline to two years after the zoledronic acid infusion.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
percentage change | -4.0 (0.8) | -4.1 (0.8) | -4.3 (1.5)

5. Secondary Outcome: Changes in Cortical Porosity Measured by High-resolution Peripheral Quantitative Computed Tomography (HR-pQCT) Scan at the Radius and Tibia From Baseline to One Year After the Zoledronic Acid Infusion.
Description: Changes in cortical porosity measured by high-resolution peripheral quantitative computed tomography (HR-pQCT) scan at the radius and tibia from baseline to one year after the zoledronic acid infusion.
Time Frame: from baseline to one year after the zoledronic acid infusion.
Population: Changes in cortical porosity at the radius from baseline to one year after the zoledronic acid infusion.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
percentage change | -2.5 (7.4) | -1.6 (6.7) | -4.2 (7.2)

6. Secondary Outcome: Changes in p-CTX From Baseline to Six Months After the Zoledronic Acid Infusion.
Description: Changes in p-CTX from baseline to six months after the zoledronic acid infusion.
Time Frame: from baseline to six months after the zoledronic acid infusion.
Population: Changes in p-CTX from baseline to six months after the zoledronic acid infusion.
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
ug/l | 0.60 (0.35) | 0.47 (0.24) | 0.47 (0.20)

7. Secondary Outcome: Changes in p-CTX From Baseline to 12 Months After the Zoledronic Acid Infusion.
Description: Changes in p-CTX from baseline to 12 months after the zoledronic acid infusion.
Time Frame: from baseline to 12 months after the zoledronic acid infusion.
Population: Changes in p-CTX from baseline to 12 months after the zoledronic acid infusion.
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
ug/l | 0.58 (0.23) | 0.40 (0.20) | 0.49 (0.21)

8. Secondary Outcome: Morphometric Vertebral Fractures Assessed by Vertebral Fracture Assessment (VFA) One and Two Years After the Zoledronic Acid Infusion.
Description: Morphometric vertebral fractures assessed by vertebral fracture assessment (VFA) one and two years after the zoledronic acid infusion.
Time Frame: one and two years after the zoledronic acid infusion.
Population: Morphometric vertebral fractures assessed by vertebral fracture assessment (VFA) two years after the zoledronic acid infusion.
Measure: Number; unit: participants
Arm/Group | 6-month Group | 9-months Group | Observation Group
Number analyzed (Participants) | 20 | 20 | 21
participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 2 - 2.5 years
Groups:
- 6-month Group: Zoledronate: administrated at baseline.
  Zoledronate re-administrated: If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site.
- 9-months Group: Zoledronate: administrated depending on increase in s-CTX (above 1.26 ug/l) or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 3.
  Zoledronate re-administrated: If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site.
- Observation Group: Zoledronate: administrated depending on increase in s-CTX (above 1.26 ug/l), decrease in BMD (more than 5% at any site), or the occurrence of an osteoporotic clinical vertebral or hip fracture, but no later than at month 6.
  Zoledronate re-administrated: If s-CTX increases above 1.26 ug/l or BMD decreases more than 5% at any site.
Arm/Group | 6-month Group | 9-months Group | Observation Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 4/21
Other Adverse Events (participants affected / at risk) | 18/20 | 18/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-month Group (N=20) | 9-months Group (N=20) | Observation Group (N=21)
Cancer (Investigations) | 0 (0) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-month Group (N=20) | 9-months Group (N=20) | Observation Group (N=21)
Flu-like symptoms after ZOL treatment (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (8) | 16 (16)
Infection (unspecified) + Musculoskeletal symptoms (Infections and infestations) | 13 (13) | 18 (18) | 15 (15)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Open-label design, no assessment by VFA or X-ray of VFx at baseline, changes in treatment not in accordance with the protocol. Information about BMD before initiation of DMAB is not available and the BMD loss can therefore not be evaluated in the context of the BMD gain during DMAB. Our p-CTX cutoff was 50% above the normal range for postmenopausal women and elderly men and it cannot be ruled out that the outcome of the study would have been different with a different cutoff.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03087851/Prot_SAP_000.pdf